CLINICAL TRIAL: NCT00238576
Title: Lamotrigine in the Treatment of Bipolar Disorder in Women of Reproductive Age
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Natalie Rasgon, Principal Investigator, Stanford University
Other Study IDs: 79890; SPO# 30264
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2012-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
This project will expand current knowledge of reproductive biology in women with bipolar disorder as well as assessing the impact of lamotrigine use for the treatment of bipolar disorder on reproductive function. Specifically, this study examines mood over the menstrual cycle and ovulation for three consecutive menstrual cycles in women treated for bipolar I, II, or NOS (not otherwise specified) with lamotrigine. In addition, testosterone and lipid concentrations will be measured before the participant starts receiving lamotrigine, as well as six months after receiving lamotrigine.

ELIGIBILITY:
Inclusion Criteria::

* Female
* Ages 18 through 45
* Diagnosis of bipolar disorder (I, II, or NOS)
* Willing to sign the Human Subject Protection Consent Form prior to enrollment into the study
* Willing to use lamotrigine
* Never used lamotrigine prior to study entry Exclusion Criteria:- Unwilling or unable to comply with study requirements, e.g. complete forms, or attend scheduled evaluations
* Significant alcohol and/or substance abuse or dependence within the prior 6 months
* Used lamotrigine prior to study entry, or currently using lamotrigine at study entry

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females age 18 through 45 with a diagnosis of bipolar, considering treatment with Lamotragine.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Changes in weight, glucose, lipid levels , insulin and testosterone concentrations over 6 months onmedication | 6 months
  This is a research study to determine how effective lamotrigine is in the treatment of bipolar disorder in women of reproductive age. Participants are between the ages of 18 and 45, have been diagnosed with bipolar disorder, and have indicated that they are about to begin or are considering treatment with lamotrigine. The purposes of this study are to explore the safety of lamotrigine in treating bipolar I disorder, bipolar II disorder, and rapid cycling bipolar disorder in women compared to other mood stabilizers and anti-depressants. In addition, this study aims to explore lamotrigine's effects on the association between the mood and the menstrual cycle and to compare the effects of various medications that participants receive for treatment of their illness in regards to reproductive hormone levels.

SECONDARY OUTCOMES:
Menstrual cycle length and presence or absence of ovulation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Natalie Rasgon, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Department of Psychiatry and Behavioral Sciences, Stanford University School of Medicine, Stanford, California
  - Stanford University School of Medicine, Stanford, California